CLINICAL TRIAL: NCT03072407
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Sequential Parallel Group, MAD Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PB-119 to Subjects With T2DM
Brief Title: MAD Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PB-119 to Subjects With T2DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP-PB119-US01-01
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: placebo-control , parallel
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PB-119 injection placebo (Placebo Comparator): totally 8 subjects will have PB-119 injection placebo once per weekly for 4 weeks.
  Interventions: Biological: PB-119 injection placebo
- PB-119 injection 25ug (Experimental): totally 8 subjects will have PB-119 injection 25 ug once per weekly for 4 weeks
  Interventions: Biological: PB-119 injection
- PB-119 injection 50ug (Experimental): totally 8 subjects will have PB-119 injection 50 ug once per weekly for 4 weeks
  Interventions: Biological: PB-119 injection
- PB-119 injection 100ug (Experimental): totally 8 subjects will have PB-119 injection 100 ug once per weekly for 4 weeks
  Interventions: Biological: PB-119 injection
- PB-119 injection 200ug (Experimental): totally 8 subjects will have PB-119 injection 200 ug once per weekly for 4 weeks
  Interventions: Biological: PB-119 injection

INTERVENTIONS:
Biological: PB-119 injection
  Arms: PB-119 injection 100ug; PB-119 injection 200ug; PB-119 injection 25ug; PB-119 injection 50ug
Biological: PB-119 injection placebo
  Arms: PB-119 injection placebo

SUMMARY:
This was a phase 1, randomized, double-blind, placebo-controlled, sequential parallel group, MAD study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of four once-weekly subcutaneous doses of PB-119 to subjects with T2DM.

DETAILED DESCRIPTION:
Dose levels of 25 µg, 50 µg, 100 µg and 200 µg with a dosing regimen of once weekly for 4 consecutive weeks will be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Patients in whom T2DM has been diagnosed for at least 3 months prior to screening and have not been taking any treatment but have made lifestyle modifications (i.e., diet and exercise) for at least 4 weeks or are taking metformin (with no change in the treatment including dose over the past 2 months).
2. In good general health as determined by the investigator at screening evaluation
3. Male and/or female subjects between the ages of 18 and 70 years, inclusive;
4. Are capable of giving informed consent and complying with study procedures;
5. Body Mass Index (BMI) of approximately 22 to 40 kg/m2;
6. Fasting C-peptide test result must be >0.4 nmol/L;
7. HbA1c ≥6.5 % and ≤12%;
8. Female subjects must have a negative urine pregnancy test result prior to enrollment.
9. Nonsmoker,
10. Willing and able to adhere to study restrictions and to be confined at the clinical research center.

Exclusion Criteria:

1. Subjects with a personal or family history of medullary thyroid carcinoma (MTC) or in subjects with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2);
2. Screening fasting blood glucose ≤100 or ≥270 mg/dL
3. Type 1 diabetes mellitus, or latent autoimmune diabetes in adults; diabetic neuropathy, retinopathy or nephropathy;
4. Previous treatment with an approved or investigational GLP-1 mimetic;
5. Patients treated with any investigational drugs within 6 weeks of screening;
6. Subjects with pancreatitis;
7. Clinically significant gastrointestinal disorder
8. History or symptoms of clinically significant cardiovascular disease, particularly coronary artery disease, arrhythmias, atrial tachycardia,
9. Uncontrolled hypertension at screening;
10. History of clinically significant central nervous system disease including: transient ischemic attack, stroke, seizure disorder, depression,
11. History of liver disease
12. History of clinically significant renal disease
13. Uncontrolled severe dyslipidemia;
14. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
15. A hospital admission or major surgery within 30 days prior to screening;
16. A history of prescription drug abuse, or illicit drug use within 6 months prior to screening;
17. A history of alcohol abuse according to medical history within 6 months prior to screening;
18. A positive screen for alcohol, or drugs of abuse;
19. An unwillingness or inability to comply with food and beverage restrictions during study participation;
20. Use of prescription or over-the-counter (OTC) medications, and herbal An
21. Unwillingness of male participants to use appropriate contraceptive measures if engaging in sexual intercourse with a female partner of childbearing potential. Appropriate measures include use of a condom and spermicide and, for female partners, use of an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, progesterone subdermal implants, or a tubal ligation. Sexual intercourse with pregnant or lactating women is prohibited

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
the number of AEs and the finding from the physical examination, the abnormal lab results | accessed up to 4 weeks
  include monitoring of AEs, vital signs (blood pressure, pulse rate, respiratory)

SECONDARY OUTCOMES:
PB-119 blood plasma concentration | accessed up to 4 weeks
  to collect PB-119 blood plasma concentration of the subjects who use PB-119 intervention
PB-119 antibody | accessed up to 4 weeks
  the number of subjects who are with positive antibody results
Insulin sensitivity (SI) | accessed up to 4 weeks
  be estimated from glucose and insulin concentration
Beta-cell Responsivity Index | accessed up to 4 weeks
  be estimated from serum glucose and c-peptide concentrations
Disposition Index | accessed up to 4 weeks
  be calculated for each individual subject as the product of SI and Φtotal

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Tracey, Dr., Principal Investigator — Frontage Clinical Services, Inc.
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Frontage Clinical Services. Inc., Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No